CLINICAL TRIAL: NCT06379048
Title: The Impact of Different Skin Suture Methods in Episiotomy Repair on Healing and Pain: A Randomized Clinical Trial
Brief Title: The Impact of Different Skin Suture Methods in Episiotomy Repair on Healing and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Emre Kar, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021.12.282
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Labor; Prolonged, Second Stage; Episiotomy Wound
Keywords: Labor; Vaginal Birth; Episiotomy; Suturing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- M-Suture (Active Comparator): Episiotomy repair is completed until the skin closure. Interrupted mattress suturing technique is applied to this arm.
  Interventions: Procedure: Mattress Suturing
- I-Suture (Active Comparator): Episiotomy repair is completed until the skin closure. Interrupted primary suturing technique is applied to this arm.
  Interventions: Procedure: Primary Suturing
- SC-Suture (Active Comparator): Episiotomy repair is completed until the skin closure. Continuous subcutaneous suturing technique is applied to this arm.
  Interventions: Procedure: Continuous Subcutaneous Suturing

INTERVENTIONS:
Procedure: Mattress Suturing — Horizontal mattress suture in interrupted fashion
  Arms: M-Suture
Procedure: Primary Suturing — Horizontal primary suture in interrupted fashion
  Arms: I-Suture
Procedure: Continuous Subcutaneous Suturing — Subcutaneous suture in continuous fashion
  Arms: SC-Suture

SUMMARY:
Episiotomy is the intentional incision of the perineum during vaginal birth in order to accelerate the active phase of labor. This study aimed to compare various skin closure techniques in episiotomy repair.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous
* Age between 18 to 45
* Given birth in our labor ward

Exclusion Criteria:

* Multiparous
* having deep vaginal lacerations
* having abnormalities in fetus
* Rheumatologic diseases
* Postpartum bleeding
* Shoulder Dystocia
* Operative Delivery
* Using antithrombotic or anticoagulant medications

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cam and Sakura City Hospital, Istanbul, Basaksehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon request for at least 2 years after publication.
Time Frame: IPD will be available upon request for at least 2 years after publication.
Access Criteria: Contact with Corresponding Author

REFERENCES:
- [Result] Yuksel S, Ustun A, Kar E, Ozcan A, Callioglu N. The impact of different skin Suture methods in episiotomy repair on healing and pain: A randomized clinical trial. Health Care Women Int. 2025;46(9):1015-1029. doi: 10.1080/07399332.2025.2499498. Epub 2025 May 5. PMID 40323943

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | M-Suture | I-Suture | SC-Suture
Started | 44 | 44 | 44
Completed | 43 | 43 | 43
Not Completed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M-Suture | I-Suture | SC-Suture | Total
Number analyzed (Participants) | 43 | 43 | 43 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.6 (2.9) | 24.9 (4.8) | 24.1 (4.1) | 23.9 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 43 | 129
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 43 | 43 | 43 | 129
Smoker [Count of Participants; unit: Participants] | 2 | 3 | 6 | 11
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 28.4 (4.5) | 27.3 (3.1) | 28.3 (5) | 28 (4.2)
Gestational Age at Delivery [Mean (Standard Deviation); unit: weeks] | 39.15 (1.5) | 38.56 (2.14) | 39.21 (1.33) | 38.97 (1.66)
Labor Induction [Count of Participants; unit: Participants] | 30 | 26 | 26 | 82
Active Birth Phase Duration (hours) [Mean (Standard Deviation); unit: hours] | 4.52 (3.89) | 4.56 (3.22) | 5.02 (3.55) | 4.7 (3.55)

OUTCOME MEASURES:

1. Primary Outcome: Healing by Redness, Edema, Ecchymosis and Discharge (REEDA) Score
Description: Healing is assessed by Redness, Edema, Ecchymosis and Discharge (REEDA) Score
  REEDA Scale:
  Healed: 0; moderately healed: 1 to 5; mildly healed: 6 to 10; and not healed: 11 to 15
Time Frame: in postpartum day 15
Measure: Median (Full Range); unit: REEDA Score
Arm/Group | M-Suture | I-Suture | SC-Suture
Number analyzed (Participants) | 43 | 43 | 43
REEDA Score | 1 [0 to 10] | 1 [0 to 9] | 0 [0 to 5]

2. Primary Outcome: Pain by Visual Analog Scale (VAS)
Description: Pain is assessed from 0 (none) to 10 (extreme) by Visual Analog Scale (VAS)
Time Frame: in postpartum day 15
Measure: Median (Full Range); unit: VAS Score
Arm/Group | M-Suture | I-Suture | SC-Suture
Number analyzed (Participants) | 43 | 43 | 43
VAS Score | 2 [0 to 10] | 2 [0 to 10] | 1 [0 to 8]

ADVERSE EVENTS:
Time Frame: 15 days
Description: Episiotomy repair is a relatively simple procedure and is not typically associated with life-threatening mortality or long-term morbidity that would significantly impact quality of life. The most significant potential morbidity is related to anal sphincter injury; however, patients with such injuries were not included in this study.
Arm/Group | M-Suture | I-Suture | SC-Suture
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 4/43 | 2/43 | 3/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M-Suture (N=43) | I-Suture (N=43) | SC-Suture (N=43)
Dehiscense (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0)
Urinary Incontinence (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 2 (2)
Fecal Incontinence (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT06379048/Prot_SAP_000.pdf